CLINICAL TRIAL: NCT04343495
Title: Pilot Studies of UV-A, UV-B, and Blue-light Dosimetry Sensors
Brief Title: UV and Bluelight Dosimetry
Status: Withdrawn | Type: Observational
Why Stopped: PI left institution and study has not begun enrollment.
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Shuai (Steve) Xu, Principal Investigator, Northwestern University
Other Study IDs: STU00209872
Record Dates: First submitted 2020-03-30; First posted 2020-04-13 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Environmental Exposure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Wearable Ultra Violet (UV) and blue-light sensors — Non-blinded

SUMMARY:
The objective of this study to assess the efficacy of wearable Ultra Violet (UV) and blue-light sensors in measuring exposure to UV radiation and blue light in a variety of environments and activity settings.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old
* Subjects willing and able to comply with requirements of the protocol
* Subjects speaking English

Exclusion Criteria:

* Age <18 years old
* Subjects unwilling and unable to comply with requirements of the protocol
* History of skin allergy to medical adhesive tape or rubber bands/elastic
* Lack of proficiency in English
* Skin disorders affecting skin integrity

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of various types of light exposure at various, targeted regions of the body while engaging in a different activities and settings. | Time Frame: 1 year
  After sensors are removed researchers will collect dosimetry data using a phone application using Near Field Communication (NFC) with a phone that is restricted to research use only in this study. Location, indoor/outdoor conditions and time that the devices are used will be recorded by the study team.
  Location, external environmental factors (weather, UV index) and activities will be recorded by the research administrators.